CLINICAL TRIAL: NCT00858897
Title: Regulation of Glutathione Homeostasis in Adolescents With Type 1 Diabetes - Study A
Brief Title: Glutathione Metabolism in Adolescents With Type 1 Diabetes - Study A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Dominique Darmaun, Physician, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: JDRF 1-2006-627-A
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Glutathione
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normoglycemia (Experimental): 80-140 mg/dL
  Interventions: Other: Cysteine isotope infusion at normoglycemia vs hyperglycemia; Drug: Regular Insulin
- Hyperglycemia (Experimental): 200-250 mg/dL
  Interventions: Other: Cysteine isotope infusion at normoglycemia vs hyperglycemia; Drug: Regular Insulin

INTERVENTIONS:
Other: Cysteine isotope infusion at normoglycemia vs hyperglycemia — L-[3,3-2H2]cysteine
Drug: Regular Insulin — Regular insulin, IV, as needed to maintain blood glucose in near-normoglycemic range (80-140 mg/dL) or hyperglycemic range (200-250 mg/mL) during metabolic studies

SUMMARY:
Glutathione is normally present at high (millimolar) levels in blood and plays an important role in the body's defense against oxidative stress, that is, against the damage caused to the body by reactive oxygen species produced by the metabolism of most nutrients, including glucose. Glutathione is a small peptide made from 3 amino acids, glutamate, cysteine, and glycine.

This study is looking at how blood sugar levels may affect the way glutathione is made and used by the body. Since glutathione is continuously synthesized and broken down, the amount of glutathione present in blood depends on the balance between its rate of synthesis and its rate of use.

In earlier studies, the investigators found that in poorly controlled diabetic teenagers, glutathione was low, not because its production was decreased, but because it was used at an excessive rate. In this study, the investigators want to determine how short-term changes in blood sugar levels affect glutathione levels. This will help improve our understanding of how diabetes affects metabolism.

DETAILED DESCRIPTION:
Adolescents with uncomplicated T1D will receive two, 5-hour infusions of deuterium-labeled cysteine on 2 separate days, a few weeks apart, while blood glucose will be maintained, using intravenous insulin infusion:

* in the hyper-glycemic range (200-250 mg/dL) on one study day, and
* near normoglycemia (80-140 mg/dL) on the other study day.

The order of the study days will be randomized.

We will determine whether the level of blood glucose at the time of study affects blood glutathione concentration, and, if so, whether this is associated with changes in the fractional rate of glutathione synthesis, as determined from the incorporation of labeled cysteine into blood glutathione over the course of the 5-hr infusion of labeled cysteine.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, using usual criteria such as: glycosuria, hyperglycemia prior to treatment
* BMI <25 kg/m2
* Age 14-18
* HbA1c>7.5%
* No evidence of diabetic complications
* Written informed consent from parents or legal guardian, and assent from patient

Exclusion Criteria:

* Presence of significant anemia (hemoglobin <11g/dL)
* Presence of intercurrent illness such as infection
* Presence of chronic disease such as other endocrine deficiency, chronic respiratory or cardiac disease
* Chronic use of medication other than insulin
* Use of vitamin or mineral supplements within 2 weeks of study

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Darmaun, MD, PhD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each of the 10 Subjects received two 5-hour intravenous infusions of L-[3,3-2H2]cysteine in the postabsorptive state on 2 separate days after blood glucose had been maintained overnight at normoglycemia or hyperglycemia, using intravenous insulin infusion. The order of the normo- and hyper-glycemia study days was randomized.
Groups:
- Normoglycemia (80-140 mg/dL), Then Hyperglycemia (200-250 mg/dL); Hyperglycemia (200-250 mg/dL), Then Normoglycemia (80-140 mg/dL): Cysteine isotope infusion at normoglycemia vs hyperglycemia: L-[3,3-2H2]cysteine on 2 separate days, in randomized order
  Regular Insulin: Regular insulin, IV, as needed to maintain blood glucose in near-normoglycemic range (80-140 mg/dL) during metabolic studies
Period: First Intervention (1 Day)
Arm/Group | Normoglycemia (80-140 mg/dL), Then Hyperglycemia (200-250 mg/dL) | Hyperglycemia (200-250 mg/dL), Then Normoglycemia (80-140 mg/dL)
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Washout (~9 Days)
Arm/Group | Normoglycemia (80-140 mg/dL), Then Hyperglycemia (200-250 mg/dL) | Hyperglycemia (200-250 mg/dL), Then Normoglycemia (80-140 mg/dL)
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: 2nd Intervention (1 Day)
Arm/Group | Normoglycemia (80-140 mg/dL), Then Hyperglycemia (200-250 mg/dL) | Hyperglycemia (200-250 mg/dL), Then Normoglycemia (80-140 mg/dL)
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects Enrolled: Adolescents with Type 1 Diabetes
Arm/Group | All Subjects Enrolled
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10
HbA1C [Mean (Standard Deviation); unit: percent of total hemoglobin] — percent of total hemoglobin, reflecting average blood glucose control over the previous 3- to 6-month period
  percent of total hemoglobin | 9.2 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Glutathione Concentration
Description: umol/L
Time Frame: Up to 30 minutes post- 5 hour infusion on Day 1 (First Intervention) and up to 30 minutes post- 5 hour infusion on Day 14 (Second Intervention)
Population: Each of the 10 Subjects received two 5-hour intravenous infusions of L-[3,3-2H2]cysteine in the postabsorptive state on 2 separate days after blood glucose had been maintained overnight at normoglycemia or hyperglycemia, using intravenous insulin infusion.
Measure: Mean (Standard Error); unit: umol/L
Groups:
- Normoglycemia (80-140 mg/dL); Hyperglycemia (200-250 mg/dL): Cysteine isotope infusion at normoglycemia vs hyperglycemia: L-[3,3-2H2]cysteine
  Regular Insulin: Regular insulin, IV, as needed to maintain blood glucose in near-normoglycemic range (80-140 mg/dL) or hyperglycemic range (200-250 mg/mL) during metabolic studies
Arm/Group | Normoglycemia (80-140 mg/dL) | Hyperglycemia (200-250 mg/dL)
Number analyzed (Participants) | 10 | 10
umol/L | 541 (232) | 551 (169)

ADVERSE EVENTS:
Groups:
- Normoglycemia (80-140 mg/dL): Cysteine isotope infusion at normoglycemia vs hyperglycemia: L-[3,3-2H2]cysteine
  Regular Insulin: Regular insulin, IV, as needed to maintain blood glucose in near-normoglycemic range (80-140 mg/dL) during metabolic studies.
  Each of the 10 Subjects received two 5-hour intravenous infusions on 2 separate days after blood glucose had been maintained overnight at normoglycemia or hyperglycemia, using intravenous insulin infusion.
- Hyperglycemia (200-250 mg/dL): Cysteine isotope infusion at normoglycemia vs hyperglycemia: L-[3,3-2H2]cysteine
  Regular Insulin: Regular insulin, IV, as needed to maintain blood glucose in hyperglycemic range (200-250 mg/mL) during metabolic studies.
  Each of the 10 Subjects received two 5-hour intravenous infusions on 2 separate days after blood glucose had been maintained overnight at normoglycemia or hyperglycemia, using intravenous insulin infusion.
Arm/Group | Normoglycemia (80-140 mg/dL) | Hyperglycemia (200-250 mg/dL)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes